CLINICAL TRIAL: NCT00491543
Title: A Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of ALT 2074 in Subjects With Type 2 Diabetes Who Have a Haptoglobin Type 2-2 Genotype and Coronary Artery Disease
Brief Title: Evaluation of ALT-2074 in Subjects With Type-2 Diabetes, Haptoglobin Type 2-2 Genotype and Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-2074-201
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2007-06

CONDITIONS: Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ALT-2074

SUMMARY:
ALT-2074 (BXT-51072) belongs to a class of drugs called "glutathione peroxidase mimics." ALT-2074 works by imitating a substance produced in various tissues in the body, which prevents damage of the heart and blood vessels. Diabetic patients with a haptoglobin 2-2 genotype have poor cardiovascular clinical outcomes.

The purpose of this study is to assess the safety, the pharmacokinetic profile and characterize the effect on biomarkers of inflammation and oxidative stress of repeat doses of ALT 2074. Subjects must be diabetic, with evidence of coronary artery disease and a haptoglobin 2-2 genotype

DETAILED DESCRIPTION:
Subjects will be male and female, 18 to 75 years old, with Type 2 diabetes mellitus, a documented or suspected history of coronary artery disease, and a Haptoglobin type 2-2 (Hp 2-2) genotype. Subjects on prescribed anti-diabetic and coronary artery disease medications may continue to take their medications throughout the study.

Subjects who qualify will receive active drug (ALT-2074 20 mg, 40 mg or 80 mg) or placebo every 8 hours for 28 days. There will be three sequential cohorts of increasing doses of active drug. There will be 2 follow-up visits (Days 35 and 42). Blood and urine tests for safety (chemistry and hematology), pharmacokinetics and relevant biomarkers to measure inflammation and oxidative stress will be performed throughout the study. Electrocardiograms and 24-hour Holter monitoring will also be performed at various time points during the study.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, 18 to 75 years of age.
2. Diagnosis of Type 2 diabetes mellitus
3. Stable coronary artery disease (CAD) documented or suspected, not requiring adjustment for ≥2 months, as determined by: a. A history of myocardial infarction verified by Q-wave electrocardiogram and/or medical records, occurring greater than 6 months before the screening Visit; OR b. A coronary angiogram and/or stress test; OR c. A ankle brachial pressure index less than 0.9; OR d. Age greater than 60 years of age
4. Hp 2-2 genotype.
5. Ability to communicate and comply with all study requirements.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-06; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Biomarkers of inflammation and oxidative stress | 28 days
Safety | 28 days
Pharmacokinetics | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey G Geohas, MD, Principal Investigator — Radiant Research; Michale Noss, MD, Principal Investigator — Radiant Reasearch
Locations (2):
- United States (2):
  - Radiant Research, Chicago, Illinois
  - Radiant Research, Cincinnati, Ohio

REFERENCES:
- [Background] Blum S, Asaf R, Guetta J, Miller-Lotan R, Asleh R, Kremer R, Levy NS, Berger FG, Aronson D, Fu X, Zhang R, Hazen SL, Levy AP. Haptoglobin genotype determines myocardial infarct size in diabetic mice. J Am Coll Cardiol. 2007 Jan 2;49(1):82-7. doi: 10.1016/j.jacc.2006.08.044. Epub 2006 Dec 13. PMID 17207726